CLINICAL TRIAL: NCT03447041
Title: Zhongshan Ophthalmic Center, Sun Yat-Sen University,China
Brief Title: Visual Quality and Contrast Sensitivity Function for Limbal Dermoid Children After Corneal Transplantation
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Yuanjin PI group, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: ZOC20171217
Record Dates: First submitted 2017-12-17; First posted 2018-02-27 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Limbal Dermoid
Keywords: Keratopathy; Visual Quality; Contrast Sensitivity Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the keratoplasty group: Patients with limbal dermoid who accepted cornea transplantation surgery after 1 year were performed quick CSF from Adaptive Sensory Technology company
- the normal group: normal children without ocular disease

SUMMARY:
This study is to inquiry the contrast sensitivity function in the 50 eyes of limbal dermoid children with keratoplasty with quick contrast sensitivity function (quick CSF) test, as well asa to analyze its relationship between visual quality.

DETAILED DESCRIPTION:
Limbal dermoid(LD) is a congenital benign tumor that consist of overgrowths of epidermal appendages that influence vision and cause visual abnormalities due to the induced corneal astigmatism. A large proportion of patients, all of whom had epibular dermoids, has amblyopia. In a previous study, keratoplasty, such as LKP (Lamellar Keratoplasty) or PKP (Penetrating Keratoplasty), was shown to facilitate the reconstruction of appearance, and improve visual acuity significantly postoperatively. However, the reestablishment of visual acuity and visual function are always ignored by parents after visual appearance recovery. Several studies have evaluated the visual acuity and objective and subjective visual function of patients after keratoplasty. These outcomes include contrast sensitivity (CS), refractive error, graft clarity, anterior and posterior corneal higher order aberration, and vision-related quality of life. Although a subjective visual function assessment has been deemed critical, postkeratoplasty patients with vision complaints are not uncommon despite clear grafts and relatively good visual acuity, and the visual function evaluation for LD were relatively less.

50 eyes of 50 limbal dermoid children with corneal transplantation more than 1 year were included in this study. All participants underwent an ophthalmic examination that included slit-lamp biomicroscopy, visual acuity, quick CSF under full optical correction, 9-SF life quality questionnaire and fundus examination. Then the normal group would be covered by the positive spherical lens of 1.0D to 6.0D to repress the BCVA to 0.1 to 0.9 respectively to compare the visual functions with the keratoplasty patients on the same visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Accept the corneal transplantation based on the clinical diagnosis of ocular surface disease;
* more than 7 and less than 60 years old;
* absence of other ocular disorders and no history of eye surgery and other systemic diseases.

Exclusion Criteria:

* less than 7 or more than 60 years old;
* with the history of eye surgery and other systemic diseases.

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There would include 50 eyes of 50 patients with corneal transplantation (the keratoplasty group) and 15 eyes of 15 normal subjects (the normal group) in this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The contrast sensitivity function tested by quick CSF in the keratoplasty group | on 1 year postkeratoplasty
  The quick CSF (contrast sensitivity function) tests including AULCSF (the area under the log CSF) and Cutoff SF (Cutoff sensitivity function)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol
Time Frame: Starting in March 2018
Access Criteria: The Visual Quality and Contrast Sensitivity Function of the keratoplasty group and the normal group

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT03447041/Prot_SAP_000.pdf